CLINICAL TRIAL: NCT00719589
Title: Outcomes of Pudendal InterStim
Status: Completed | Type: Observational
Sponsor: Corewell Health East (Other)
Responsible Party: Kenneth Peters, MD, William Beaumont Hospital-Royal Oak
Other Study IDs: 2008-152
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2010-03

CONDITIONS: Voiding Dysfunction
Keywords: Voiding Dysfunction; Interstim

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patient who have had implantation of an interstim.

SUMMARY:
The purpose of this study is to determine how many patients who have failed treatment with a sacral lead can achieve good results with a pudendal, patients satisfaction with the results of each lead, complication rates after pudendal lead placement, and how many patients have required reprogramming of their device with EMG testing( a more costly procedure).

DETAILED DESCRIPTION:
InterStim is a bladder pacemaker device that has been in use for over 10 years for patients with voiding dysfunction. Although standard of care is to place the lead at the sacral nerve, in some patients a better response is obtained by placing the lead at the pudendal nerve.

Data will be collected from the subjects medical records and a questionnaire will be mailed one time to assess patients perception of improvement and treatment satisfaction after pudendal Interstim.

ELIGIBILITY:
Inclusion Criteria:

* All patients having had Interstim with a pudendal lead at Beaumont

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at William Beaumont Hospital-Royal Oak who have had implantation of an Interstim with a pudendal lead.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2008-07; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
To determine the outcomes of pudendal interstim in terms of number of failed sacral lead patients that can be salvaged with a pudendal lead, | 2 years

SECONDARY OUTCOMES:
To determine the outcomes of pudendal interstim in terms of complications | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth M Peters, MD, Principal Investigator — William Beaumont Hospital - Royal Oak
Locations (1):
- William Beaumont Hospital-Royal Oak, Royal Oak, Michigan, United States